CLINICAL TRIAL: NCT00668928
Title: Effect of Dietary Polyphenols on Insulin Sensitivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: David J. Baer, ARS/USDA/BHNRC
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-252
Record Dates: First submitted 2008-04-23; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Polyphenols (flavon-3-ol monomers and oligomers) — Flavanols

SUMMARY:
A large and growing segment of the population is prediabetic. Dietary interventions that improve insulin sensitivity may be important in preventing the progression to full-blown diabetes in these individuals. Foods and dietary compounds that increase insulin sensitivity are likely to help maintain a healthier body composition. This pilot study will provide data to evaluate the role of dietary plant polyphenols in improving insulin sensitivity.

DETAILED DESCRIPTION:
How does the amount consumed of cocoa and tea polyphenols (flavon-3-ol monomers and oligomers) affect insulin sensitivity in insulin resistant individuals?

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are insulin resistant based on routine clinical measurements (Stern et al., 2005).

Exclusion Criteria:

* BMI < 27 kg/m²
* Age < 25 and > 65 years
* Pregnant women or women who plan on becoming pregnant during the study
* Postpartum women
* Lactating women
* Diabetes mellitus
* Kidney disease
* Liver disease
* Certain cancers
* Smokers

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, PhD, Principal Investigator — ARS/USDA/BHNRC